CLINICAL TRIAL: NCT02775305
Title: The Effects of Frailty on Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cynthia Delgado, Staff Physician, San Francisco Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IK2CX000527 (NIH)
Record Dates: First submitted 2014-12-12; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Sarcopenia; Chronic Kidney Disease
MeSH Terms: conditions — Sarcopenia; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Not frail (No Intervention): Source of these participants will be the same as those who screen into the study; patients with chronic kidney disease receiving care at the San Francisco Veteran Affairs Medical Center. Based on initial screening if participants do not meet criteria for frailty, baseline screening data will be used for comparative analysis as the no intervention arm.
- Frail (Experimental): Source of these participants will be the same as those who screen into the study; patients with chronic kidney disease receiving care at the San Francisco Veteran Affairs Medical Center. Based on initial screening if participants meet criteria for frailty participants will be enrolled in the intervention arm. Participants who are ambulatory regardless of co-morbidities will not be excluded from the study.
  Interventions: Behavioral: Frail

INTERVENTIONS:
Behavioral: Frail — Slowness/weakness: Physical therapy(PT) strength and gait training. A standardized strengthening program will be prescribed, to be performed at home. Additional in-person PT training will be provided to those who are severely deconditioned .
  Weight loss/malnutrition: A licensed nutritionist specializing in kidney disease will meet with participants for 3 one-hour one-on-one nutritional counseling.
  Low physical activity: Participants will receive individualized walking recommendations using a pedometer. Walking activity will be assessed weekly, and new goals for increasing steps in the following week will be set.
  Exhaustion: Those who meet criteria for severe depression using the center for epidemiologic studies depression (CES-D) scale will be immediately referred to psychiatry for counseling for patient safety. All others will participate in cognitive behavioral coping techniques.
  Arms: Frail

SUMMARY:
Frailty is a syndrome characterized by decreased reserve and diminished resistance to stressors. The proposed research will evaluate the association of frailty with chronic kidney disease (CKD). The prevalence of frailty increases with age and with CKD, but studies are needed to determine whether frailty is associated with worsening of CKD and whether intervention to treat frailty can improve physical functioning and health-related quality of life (HRQOL) as well as slow progression of CKD.

DETAILED DESCRIPTION:
The intervention is a 6-month prospective interventional pilot study targeted to each domain of frailty. Subjects will be screened into the study by testing each domain; only those who meet criteria for frailty will be included in the study. The clinical intervention, which all subjects will receive, will begin immediately upon enrollment and completion of baseline measurements. Upon enrollment the 3 most recent previous outpatient serum creatinine measurements (up to 1 year) will be used to determine baseline slope of estimated glomerular filtration rate (eGFR). The main objectives of the pilot study will be to gain knowledge in the successful implementation and completion of an intervention targeted toward frailty. Ultimately information ascertained from this pilot will serve as a springboard for planning of a randomized trial aimed at addressing all the domains of frailty, which is key given that previous studies have only implemented interventions aimed at a single domain or in pairs, but no studies have evaluated the extent to which frailty can be reversed through a cohesive intervention addressing all domains together. The intervention outlined in this proposal is comprehensive and focused while maintaining feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease Stage III to IV
* Receiving care at the San Francisco Veterans Affairs Medical Center
* Able to consent in English

Exclusion Criteria:

* Early chronic kidney disease
* individuals with acute kidney injury
* non-ambulatory

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Pedometer Step Count | Change from baseline step count to 6 months
  The number of steps achieved over the 6 month period will be assessed. Pedometer data is collected each week. Based on the weekly achieved counts a new goal is generated for each participant. This assessment will include study investigators collecting step count logs from the participant on a weekly basis.
Physical Function | baseline and 6 months
  Change in physical functioning will be assessed using the short physical performance battery (SPPB). Investigators will compare baseline Short physical performance battery (SPPB) score to 6 month score to determine change in functioning as a result of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Delgado, MD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- Department of Veterans' Affairs Medical Center, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.